CLINICAL TRIAL: NCT06823804
Title: Research and Monitoring of Ventilation-Perfusion Imaging Technology Using Electrical Impedance Tomography for ARDS Patients' PEEP Trial Lung Ventilation Strategies Clinical Study.
Brief Title: Impact of PEEP Trials on Ventilation-Perfusion Matching in ARDS Patients
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022325
Record Dates: First submitted 2024-12-25; First posted 2025-02-12 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2024-12

CONDITIONS: ARDS
Keywords: ventilation/perfusion ratio; Electrical impedance tomography; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Observational study、Exploratory research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- evaluate the feasibility of using EIT to calculate regional recruitment-to-inflation (R/I) ratios (Experimental): Regional R/I ratios were computed for the global lung, dorsal (dependent), and ventral (non-dependent) regions of interest (ROIs), which were defined as 50% of the ventro-dorsal lung diameter based on EIT imaging.compare the predictive value of regional (dorsal and ventral) versus global R/I for recruitment success in moderate-severe ARDS.
  Interventions: Drug: 10ml of 10% saline is injected centrally

INTERVENTIONS:
Drug: 10ml of 10% saline is injected centrally — The first phase of the study is an observational study that does not alter the clinical treatment plan.
  The experimental group standardized PEEP step maneuver from 5 → 15 cmH₂O, maintained for 3 minutes. Continuous EIT monitoring of regional compliance, oxygenation, hemodynamics. Dynamic strain cutoff (>0.6) or adverse events terminate the maneuver.
  Ventilation mode: volume control, tidal volume 4-6 mL/kg predicted body weight, plateau ≤28-30 cmH₂O, FiO₂ titrated for SpO₂ 88-92%.
  Other Names: Electrical impedance tomography

SUMMARY:
In the treatment of critically ill patients, mechanical ventilation is a key link, and appropriate mechanical ventilation strategies can open the alveoli and improve oxygenation, while inappropriate mechanical ventilation can increase lung injury and seriously affect the prognosis. Ventilator-related lung injury is mainly concentrated in barotrauma, volumetric injury, shear injury, and biological injury, and the monitoring of respiratory ventilation to the level of local ventilation can help to better assess the state of alveolar opening and alveolar collapse, and help to understand the uniformity of gas distribution in the lungs, which is closely related to lung injury. However, how to achieve simple, bedside and real-time lung ventilation and lung volume assessment in clinical work has always been a difficult problem to be overcome. This study intends to explore the changes of local ventilation and blood flow in the lungs during PEEP trail in patients with ARDS monitored by EIT.

DETAILED DESCRIPTION:
1. Background and Rationale ARDS is associated with heterogeneous lung collapse. The recruitment-to inflation (R/I) ratio has emerged as an index of recruitability, but is usually assessed globally. Electrical impedance tomography (EIT) enables regional assessment of ventilation and may provide more precise determinations of recruitable lung regions, particularly dorsal areas.
2. Objectives Primary objective: To compare the predictive value of regional (dorsal and ventral) versus global R/I for recruitment success in moderate-severe ARDS. Secondary objectives: To classify recruitment phenotypes and evaluate associations with oxygenation, compliance improvement, ventilator-free days, ICU length of stay, and 28-day mortality.
3. Study Design Prospective, single-centre observational cohort study in ICU patients with moderate-severe ARDS. All eligible patients undergo standardised recruitment maneuver and EIT monitoring.
4. Study Setting Ruijin Hospital, Shanghai Jiao Tong University School of Medicine ICU, December 2022 - December 2024.
5. Intervention Standardized PEEP step maneuver from 5 → 15 cmH₂O, maintained for 3 minutes. Continuous EIT monitoring of regional compliance, oxygenation, hemodynamics. Dynamic strain cutoff (>0.6) or adverse events terminate the maneuver. Ventilation mode: volume control, tidal volume 4-6 mL/kg predicted body weight, plateau ≤28-30 cmH₂O, FiO₂ titrated for SpO₂ 88-92%.
6. Measurements EIT-derived ΔEELI in dorsal and ventral regions Regional and global compliance (Crec and Crs) R/I calculated: Crec/Crs at baseline PEEP Airway opening pressure by low-flow inflation method Primary outcome: recruitment success (≥10% compliance improvement + ≥20 mmHg PaO₂/FiO₂ increase) Secondary: ventilator-free days, ICU LOS, 28-day mortality, dynamic strain
7. Statistical Analysis Plan Distribution check by Shapiro-Wilk. Paired tests for within-patient comparisons. ROC curves and Youden index for cut-off selection. Multivariate regression for mortality risk factors. Bonferroni correction for multiple comparisons.
8. Safety Monitoring Terminate RM if: MAP <65 mmHg, SpO₂ <88%, arrhythmia onset, dynamic strain >0.6.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the Berlin definition of ARDS and have been treated with mechanical ventilation (clinical diagnosis of ARDS by the attending ICU physician)
* PaO₂/FiO₂ ≤150 mmHg

Exclusion Criteria:

* Age< 18 or >90 years
* Pneumothorax, pneumomediastinum
* Hemodynamic instability (rising vasopressor need in <6h)
* Contraindications to RM or EIT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | From enrollment to the end of treatment at 28 days
  Statistical analysis of 28-day mortality
recruitment success percent | From enrollment to the end of treatment at 7 days
  recruitment( ≥10% compliance improvement ) and Re-check the blood gas ≥20 mmHg PaO₂/FiO₂ increase mean success
Correlation between EIT-derived parameters and clinical outcomes | From enrollment to the end of treatment at 28-day
  Correlation analysis between EIT-derived parameters [e.g., GI index (100%), ROI (100%), V/Q ratio, percentage of dead space (100%)] and clinical outcomes[e.g., 28-day mortality]
Change in Sequential Organ Failure Assessment (SOFA) score from baseline to day 7 | From enrollment to the end of treatment at 7 days
  Change in Sequential Organ Failure Assessment (SOFA) score from baseline to day 7
Duration of mechanical ventilation from enrollment to successful weaning | From enrollment to the end of treatment at 7 days
  Duration of mechanical ventilation in days from enrollment to successful weaning
Improvements in lung compliance | through study completion, an average of 3 month
  Change in lung compliance measured by EIT and Ventilator (C=△V/△P)during PEEP trials from baseline to 30 minutes at each PEEP level (0，5, 10, 15 and 20 cmH2O)
Regional and global compliance (Crec and Crs) | through study completion, an average of 3 month
  The EIT detection calculates the corresponding results through a continuous monitoring process that lasts approximately 3 minutes.

SECONDARY OUTCOMES:
Changes in regional ventilation-perfusion matching during PEEP trials | From enrollment to the end of treatment at 7 days
  Change in ventilation-perfusion ratio measured by EIT during PEEP trials from baseline to 30 minutes at each PEEP level (5 → 15 cmH₂O )
Change in PaO2/FiO2 ratio | From enrollment to the end of treatment at 7 days
  Change in PaO2/FiO2 ratio from baseline to day 7 measured by arterial blood gas analysis
Change in dyspnea severity | From enrollment to the end of treatment at 7 days
  Change in dyspnea severity from baseline to day 7 measured by Visual Analog Scale (VAS) score (range 0-100)
Length of ICU stay | From enrollment to the end of treatment at 7 days
  Length of ICU stay in days
Incidence of adverse events | From enrollment to the end of treatment at 7 days
  Incidence of adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0

OTHER OUTCOMES:
Change in IL-6/IL-10 ratio | From enrollment to the end of treatment at 5 days
  Change in IL-6/IL-10 ratio from baseline to day 5 measured by immunoassay
Percentage of patients achieving ventilator-free days | From enrollment to the end of treatment at 7 days
  Percentage of patients achieving ventilator-free days
Hospital costs during ICU stay | From enrollment to the end of treatment at 7 days
  Hospital costs in USD during ICU stay
Quality of life score at discharge | From enrollment to the end of treatment at 28 days
  Quality of life score at discharge measured by EQ-5D-5L instrument (range 0-1)

CONTACTS AND LOCATIONS:
Overall Officials: Hongping Qu, Study Chair — Department of Critical Care Medicine，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine; Jialin Liu, Principal Investigator — Department of Geriatrics，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine; rui zhang, Study Director — Department of Critical Care Medicine，Ruijin Hospital
Locations (1):
- Department of Critical Care Medicine，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine，Shanghai，China., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No